CLINICAL TRIAL: NCT01594060
Title: A Randomized, Comparative Study of Basal-bolus Insulin Versus Conventional Sliding-scale Regular Insulin Therapy in Management of Non-critically Ill Patients Hospitalized in the Medical Ward.
Brief Title: Basal Bolus vs. Sliding Scale for Treatment of Diabetic Patients in Medical Wards
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0042-12-EMC
Record Dates: First submitted 2012-05-07; First posted 2012-05-08 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2016-09

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin; insulin glulisine; Insulin Glargine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sliding scale (Active Comparator)
  Interventions: Drug: Insulin, regular - act rapid
- basal bolus (Active Comparator)
  Interventions: Drug: Insulin glulisine, Insulin glargine

INTERVENTIONS:
Drug: Insulin, regular - act rapid — 4 shots of regular insulin: 3 before meals and one at bedtime.
  Arms: sliding scale
Drug: Insulin glulisine, Insulin glargine — 1 shot glargine at bedtime 3 shots glulisine before meals
  Arms: basal bolus

SUMMARY:
A comparison of two treatment approaches for hyperglycemia in diabetic patients hospitalized in the medical department. The first approach is called basal-bolus in which 4 insulin shots are given daily ( 3 short acting before meals and one long acting before bed time). The second approach is called sliding scale in which short acting insulin alone is given before meals and before bed time according to the patient's glucose values. The aim is to keep fasting glucose between 140-180 mg/dl.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to internal medicine ward with blood glucose (BG) between 140-400 mg/dl.
* Known history (>6months) of diabetes.
* Aged 18-80 years old.
* Previous therapy including either diet alone or any combination of oral hypoglycemia agents, glucagon-like peptide 1 (GLP-1) analogs and long acting insulin analogs or Neutral Protamine Hagedorn (NPH).

Exclusion Criteria:

* Pregnancy
* Patients with ketoacidosis
* Patients with unknown history of diabetes
* Patients with type 1 diabetes mellitus
* Patients with clinically relevant hepatic disease or renal impairment ( serum creatinine≥2.5 mg/dl)
* Use of corticosteroid therapy
* Patient with any mental disorder preventing him to cooperate and give informed consent.
* Patients on multiple daily doses of insulin regimen.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2012-06; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)